EVALUATION OF SSS 1

## **Study Protocol for:**

**Development and Pilot Trial of an Intervention to Reduce Disclosure Recipients Negative Social** 

**Reactions and Victims Psychological Distress and Problem Drinking** 

NCT03488927

Last approved August 25, 2020

**Contents:** 

**Study Protocol** 

EVALUATION OF SSS 2

## **Research Design**

Participants were assigned to either the treatment condition or the wait-list control condition. Because a large number of participants (n = 531; 63.50% of participants invited) who were assigned to the treatment condition did not attend the actual intervention, we created three groups for the purposes of analyses: control (n = 432), treatment attender (Tx-Attender; n = 305), treatment non-attender (Tx-Nonattender; n = 531).

## **Procedures**

The study took place at a residential, medium-size public university in the northeastern United States and received approval from the university's Institutional Review Board. The university's Dean of students sent emails to randomly selected, full-time, undergraduate students between the ages of 18 and 24 on the behalf of the researchers. These emails (initial and two reminders) were sent via mass email to 7,000 students in four batches across four weeks in the fall of 2018. We also sent an email from the research team to all professors at the University with classes greater than 60 students (n = 205 professors), as identified by the course catalog. Lastly, we posted fliers in residence halls and other shared spaces about the study.

Overall, 1,831 students started the baseline survey, of whom 1,268 consented to and completed the survey. Of our final 1,268 participants, 78.4% (n = 994) were recruited via official email from the Dean of students, 14.4% (n = 183) were recruited via a friend (i.e., a friend forwarded the study information), 4.9% (n = 62) were recruited via professors, 1.3% (n = 16) were recruited via fliers, 0.6% (n = 8) were recruited via the website, and 0.4% (n = 5) were recruited in another way (e.g., "Facebook"). Qualtrics randomized participants into intervention and control groups. Participants were initially randomized at a 50/50 rate to the intervention and control conditions. However, we found that rates of intervention attendance were lower than

EVALUATION OF SSS 3

expected. Thus, in order to achieve desired numbers of intervention participants, when we reached over 400 in the control group, we began assigning 100% of participants who were randomly selected to be emailed to the intervention group. Because participants were recruited via professors and fliers were not randomly selected, these participants were randomized 50/50. Thus, 65.9% of participants were assigned to the intervention (n = 836) and 34.1% were assigned to control (n = 432). Participants randomized into the intervention group were invited to attend the intervention, which was conducted in two sessions (initial session and booster session). Initial session attendance was 36.2% (n = 303); of those, 83.1% (n = 252) attended the booster.

Participants first completed the baseline survey (Time 1). An average of two weeks later, those in the intervention group participated in the first intervention session. The follow-up survey (Time 2) occurred 6 months after the first intervention session, and, for control participants, 6 months and 2 weeks after their baseline survey (to ensure receipt of email at times comparable to intervention participants). We sent participants up to eight total text, email, and call reminders to remind them of the Time 2 survey. Of the 1,268 baseline participants, 70.1% (n = 889) completed the Time 2 survey, including 314 in the control condition and 575 in the intervention group. Participants received \$15 and \$25 gift cards for completing Time 1 and 2, respectively. Of the 305 participants who attended the first session, 252 (82.6%) attended the booster session. Participants also received reminder texts, emails, and calls to remind them about the initial and booster sessions; they received up to five of these reminders.